CLINICAL TRIAL: NCT05224843
Title: The Feasibility of the VOICES Digital Health Tool for Elder Mistreatment Screening in the Primary Care Setting (VOICES-PC Feasibility)
Brief Title: Feasibility of VOICES Elder Abuse Intervention in Primary Care Setting (VOICES-PC Feasibility)
Acronym: VOICES-PC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2000023799_b; 1R01AG060084-01 (NIH)
Record Dates: First submitted 2022-01-25; First posted 2022-02-04 (Actual); Results first posted 2023-07-17 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: Elder Abuse
MeSH Terms: interventions — Voice

STUDY DESIGN:
Intervention Model Description: VOICES Elder Abuse Intervention
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Older adults in Primary Care setting (Experimental): Elder mistreatment in the Primary Care setting.
  Interventions: Behavioral: Virtual cOaching in making Informed Choices on Elder Mistreatment Self-Disclosure (VOICES)

INTERVENTIONS:
Behavioral: Virtual cOaching in making Informed Choices on Elder Mistreatment Self-Disclosure (VOICES) — Virtual cOaching in making Informed Choices on Elder Mistreatment Self-Disclosure (VOICES) screening tool.

SUMMARY:
To test an interactive intervention to screen for Elder Abuse and Mistreatment (EM) in the Primary Care (PC) setting to promote self-identification and self-disclosure of EM.

DETAILED DESCRIPTION:
The aim of this study is to perform a feasibility evaluation (N=80) of the VOICES screening tool among older adults in the primary care setting. If VOICES is feasible for identifying suspicion of EM in primary care setting, then it will be able to connect more victims of EM to necessary services and potentially prevent a multitude of poor EM outcomes

ELIGIBILITY:
Inclusion Criteria:

* Age 60 years or older
* Alert and oriented to person and place
* Abbreviated Mental Test (AMT-4) score of 4
* Able to consent and communicate in English
* Agrees and able to use the iPad

Exclusion Criteria:

* subjects who live in nursing homes or other long-term care sitting and do not reside in community setting
* patients will be excluded if they cannot safely undergo the studies required for participation
* subjects with clear signs of EM
* Patient or clinician refusal to participate
* severe hearing and vision impairment
* COVID-19 positive

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-12-17 (Actual); Primary Completion 2022-06-22 (Actual); Study Completion 2022-06-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fuad Abujarad, PhD,MSc, Principal Investigator — Yale University
Locations (1):
- Yale Internal Medicine Associates, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Older Adults Enrolled in the Study: The number of eligible older adults who were enrolled in the VOICES study.
Period: Overall Study
Arm/Group | Older Adults Enrolled in the Study
Started | 80
Completed | 80
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Older Adults in Primary Care Setting: The number of eligible older adults enrolled in the Virtual cOaching in making Informed Choices on Elder Mistreatment Self-Disclosure (VOICES) study in the primary care setting.
Arm/Group | Older Adults in Primary Care Setting
Number analyzed (Participants) | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.1 (7.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49
  Male | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 76
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 13
  White | 66
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 80
Education [Count of Participants; unit: Participants]
  High School not Completed | 3
  High School Graduate or GED | 10
  Some college or associate's degree program | 14
  Associate's Degree | 7
  College degree (bachelor's program) | 9
  Graduate degree (master's program) | 26
  Doctorate or professional degree | 11
Household Income [Count of Participants; unit: Participants]
  Less than 25k | 11
  Between 25k to 34k | 3
  Between 35k to 49k | 3
  Between 50k to 74k | 15
  Between 75k to 99k | 6
  Between 100k to 149k | 14
  More than 150k | 15
  Refused/Unknown | 13
Marital Status [Count of Participants; unit: Participants]
  Single or Never Married | 11
  Widowed | 8
  Married or Co-habituating | 45
  Divorced | 13
  Separated | 3
  Other | 0
  Refused/Unknown | 0
Employment Status [Count of Participants; unit: Participants]
  Retired/Not Employed | 61
  Part-time | 6
  Full-time | 13
Living Arrangement [Count of Participants; unit: Participants]
  In my home | 74
  In someone else's home | 2
  Assisted living | 4
Number of Household Members [Median (Standard Deviation); unit: persons] — Population: This is based off of those who do not live alone (N=53) out of the 80 participants who completed VOICES.
  persons
    number analyzed (Participants) | 53
    (all) | 2 (0.84)
Internet Usage [Count of Participants; unit: Participants]
  Every Day | 63
  1-2 Times a Week | 4
  1-2 Times a Month | 2
  Rarely | 11
Confidence in Using Technology [Mean (Standard Deviation); unit: units on a scale] — Confidence in Using Technology is measured by a question that uses a scale of 1-10 (0= Not confident at all, 10= Very confident), where a higher score indicates greater confidence.
  units on a scale | 6.74 (2.83)
Has Living Will [Count of Participants; unit: Participants]
  Yes | 45
  No | 30
  Unknown | 5
Veteran Status [Count of Participants; unit: Participants]
  Yes | 10
  No | 70
Has Health Care Assistant [Count of Participants; unit: Participants]
  Yes | 71
  No | 6
  Unknown | 3

OUTCOME MEASURES:

1. Primary Outcome: Participation
Description: Participation will be determined by the number of patients enrolled in VOICES. Successful enrollment of 80 older adults (N=80).
Time Frame: 5-10 minutes before VOICES intervention use.
Measure: Count of Participants; unit: Participants
Groups:
- Older Adults Approached for the Study: The number of older adults approached for the study in the primary care setting.
Arm/Group | Older Adults Approached for the Study
Number analyzed (Participants) | 97
Participants | 80
Statistical Analysis 1: Comparison: Older Adults Approached for the Study; Test type: Other; Percentage of enrolled from eligible = 82.5, 95% CI 2-sided [73.7 to 88.8]

2. Primary Outcome: Usage
Description: Usage will be determined by the number of patients enrolled in the study that complete the VOICES tool. Our target is to enroll 80 older adults (N=80).
Time Frame: 5-10 minutes directly following VOICES intervention.
Measure: Count of Participants; unit: Participants
Groups:
- Older Adults Enrolled in the Study: The number of eligible older adults who were enrolled in the VOICES study in the primary care setting.
Arm/Group | Older Adults Enrolled in the Study
Number analyzed (Participants) | 80
Participants | 80
Statistical Analysis 1: Comparison: Older Adults Enrolled in the Study; Test type: Other; Percentage of enrolled from eligible = 100, 95% CI 2-sided [95.4 to 100]

3. Other Pre Specified Outcome: Acceptability
Description: Participant satisfaction will be measured using post-use satisfaction survey. Responses will be measured via two 5-point Likert scales where generally higher values represent better outcomes:
  Scale 1- Satisfaction: Where 1= "Very Dissatisfied", 2= "Dissatisfied", 3= "Neutral", 4= "Satisfied", and 5= "Very Satisfied".
  Scale 2- Agreement: Where 1= "Strongly Disagree", 2= "Disagree", 3= "Neutral", 4= "Agree", and and 5= "Strongly Agree".
Time Frame: 5-10 minutes directly following VOICES intervention use.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Older Adults in Primary Care Setting: The number of eligible older adults enrolled in the VOICES study in the primary care setting.
Arm/Group | Older Adults in Primary Care Setting
Number analyzed (Participants) | 80
units on a scale
  Level of confidentiality and privacy provided while using VOICES (Scale 1) | 4.45 (0.96)
  The time it took to complete using the VOICES tool (Scale 1) | 4.67 (0.69)
  Ability to complete VOICES on their own on the iPad, without staff assistance (Scale 1) | 4.60 (0.74)
  Time to complete the tool on the iPad was short (Scale 2) | 4.42 (0.82)
  Participant felt engaged in the tool throughout the process (Scale 2) | 4.29 (0.96)
  Audio and visual aids of the tool were helpful (Scale 2) | 4.15 (0.98)
  Participant felt fonts, size and colors of text in the tool were appropriate and readable (Scale 2) | 4.64 (0.72)
  Using this tool on the iPad was very easy (Scale 2) | 4.71 (0.66)
  I was comfortable answering questions on the iPad (Scale 2) | 4.75 (0.61)
  Using the iPad and the headphones provided more privacy (Scale 2) | 4.41 (0.84)
  Participant feels comfortable discussing mistreatment with a doctor or medical professional (Scale2) | 4.46 (0.78)
  VOICES is appropriate for learning about mistreatment (Scale 2) | 4.54 (0.67)
  VOICES is appropriate to be used in primary care setting (Scale 2) | 4.11 (1.06)
  The participant was able to complete VOICES on the iPad on their own (Scale 2) | 4.54 (0.83)
  Using VOICES on the iPad was a frustrating experience (Scale 2) | 1.74 (1.10)
  The instructions provided by VOICES digital coach were clear and easy to follow (Scale 2) | 4.70 (0.56)
  Participant confidence understanding mistreatment and resources after using VOICES (Scale 2) | 4.41 (0.85)
  Participant feels safer after using VOICES on the iPad (Scale 2) | 3.80 (1.08)
  The participant learned new, useful things about elder mistreatment (Scale 2) | 4.05 (0.98)
  Participant would like to see VOICES used by others in the community (ie. doctor's office) (Scale 2) | 4.47 (0.76)

4. Other Pre Specified Outcome: Demand
Description: Demand will be assess through examining how likely will VOICES be used by patients. To do this, the size of target population of elder mistreatment (EM) victims in the Primary Care setting will be measured by the percent who screen positive for EM and the percent who receive the Brief Negotiation Interview (BNI) portion of VOICES. The BNI is a method designed to enhance identifying EM among older adults-- the process intends to encourage reflection of the user with their behaviors and whether they are willing to seek change by identifying with and reporting their abuse.
Time Frame: 5-10 minutes directly following VOICES intervention use.
Measure: Count of Participants; unit: Participants
Arm/Group | Older Adults in Primary Care Setting
Number analyzed (Participants) | 80
Participants
  Participants who screened positive for suspicion of elder mistreatment | 6
  Participants who self-identified with elder mistreatment | 3
  Participants who self-reported elder mistreatment | 3
  Participants who received the Brief Negotiated Interview (BNI) pathway | 4
Statistical Analysis 1: Comparison: Older Adults in Primary Care Setting; Test type: Other; Percentage screened positive for EM = 7.5, 95% CI 2-sided [3.5 to 15.4]

5. Other Pre Specified Outcome: Practicality
Description: Practicality will be assessed by observing the ease of VOICES use by patients. To do this, a series of steps will be watched to determine the efficiency of implementation measured by the average time (1) to consent & orient participants to the tool and (2) needed to complete VOICES documented by the Research Assistant; and (3) patients perceived time of VOICES as measured on post-survey. Each of these will be reported as part of the overall outcome.
Time Frame: Actual time duration is assessed during VOICES use by the computer program (the actual duration of the patient's time using VOICES). Estimation of completed time is completed 5-10 minutes directly following VOICES intervention use.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Older Adults in Primary Care Setting
Number analyzed (Participants) | 80
minutes
  Actual VOICES Duration | 9.31 (4.33)
  Actual Consent Duration | 14.09 (4.54)
  Participant estimated time to completion | 18.38 (11.55)

6. Other Pre Specified Outcome: Efficacy of the Brief Negotiation Interview
Description: To look at how many patients changed their readiness to disclose after completing the Brief Negotiation Interview (BNI)
Time Frame: Measure collected 5-10 minutes directly following VOICES intervention.
Measure: Count of Participants; unit: Participants
Groups:
- Older Adults Who Accessed Brief Negotiation Interview (BNI): The number of enrolled older adults who accessed the optional Brief Negotiation Interview (BNI) pathway in the VOICES program.
Arm/Group | Older Adults Who Accessed Brief Negotiation Interview (BNI)
Number analyzed (Participants) | 4
Participants | 1
Statistical Analysis 1: Comparison: Older Adults Who Accessed Brief Negotiation Interview (BNI); Test type: Other; Percentage who changed after BNI = 25, 95% CI 2-sided [4.6 to 69.9]

7. Other Pre Specified Outcome: Accuracy
Description: To understand the accuracy of the VOICES tool, a preliminary evaluation of the accuracy of VOICES as a screening tool in correctly classifying elder mistreatment (EM) cases that were referred to Adult Protective Services (APS). The percent correct classification will be reported.
Time Frame: Measure collected up to directly following VOICES intervention to 1 week following VOICES intervention.
Population: The number of participants who used VOICES to completion and screened positive for suspicion of elder mistreatment (n=6).
Measure: Count of Participants; unit: Participants
Groups:
- Older Adults in Primary Care Setting: Enrolled older adults in the primary care setting who participated in the VOICES study.
Arm/Group | Older Adults in Primary Care Setting
Number analyzed (Participants) | 6
Participants
  Participants substantiated for elder mistreatment by the social worker | 6
  Participants referred to APS by the social worker | 1
  Cases referred to APS that were substantiated and opened: number analyzed (Participants) | 1
  Cases referred to APS that were substantiated and opened | 1
Statistical Analysis 1: Comparison: Older Adults in Primary Care Setting; Test type: Other; Percentage reported APS from EM positive = 20, 95% CI 2-sided [3.6 to 62.4]

ADVERSE EVENTS:
Time Frame: Adverse event data for each participant was collected immediately upon occurrence during their study session (approximately 5-15 minutes including post-survey activities). Overall data were collected over the entire enrollment period, from 12/15/2022 to 6/22/2022, a period of 7 months
Arm/Group | Older Adults in Primary Care Setting
All-Cause Mortality (participants affected / at risk) | 0/80
Serious Adverse Events (participants affected / at risk) | 0/80
Other Adverse Events (participants affected / at risk) | 0/80

LIMITATIONS AND CAVEATS:
This study was limited to English-speaking older adults, leading to less representation with the Hispanic/Latino population.

Providers, nurses and other clinical staff were not included in the study and outcomes only extend to older adult patients in the primary care setting.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2022-02-08): https://cdn.clinicaltrials.gov/large-docs/43/NCT05224843/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-16): https://cdn.clinicaltrials.gov/large-docs/43/NCT05224843/SAP_001.pdf
  • Informed Consent Form (2022-01-04): https://cdn.clinicaltrials.gov/large-docs/43/NCT05224843/ICF_002.pdf